CLINICAL TRIAL: NCT05167357
Title: Multicentric Evaluation of the Impact on Hypoxia Sensitivity of Patients With COVID-19
Brief Title: Coronaltitude - Multicentric Evaluation of the Impact on Hypoxia Sensitivity of Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Formation et de Recherche en Médecine de Montagne (Other)
Collaborators: University of Paris 13 (Other); Ecole Nationale des Sports de Montagne (Other)
Responsible Party: Principal Investigator, Lecoq James François, Medical Doctor, PhD. Chef de pôle urgence et médecine de montagne, Institut de Formation et de Recherche en Médecine de Montagne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CORONALTITUDE2021
Record Dates: First submitted 2021-09-05; First posted 2021-12-22 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Covid19; SARS-CoV2 Infection; Hypoxia, Altitude
Keywords: Hypoxia, high Altitude; Cardiorespiratory injury; Respiratory Tract Infections; Neurological injury; Neurotropism; Acclimatization; High Altitude Effects; High Altitude Illness; Cardiorespiratory Exercise Test; Covid19; SARS-CoV-2; Hypoxia sensibility; Hypoxic response; Carotid bodies; Chemosensitivity; Covid19, pathophysiology; hypoxia at exercise; hypoxic cardiac response at exercise; hypoxic ventilatory response at exercise
MeSH Terms: conditions — COVID-19; Altitude Sickness; Hypoxia; Respiratory Tract Infections; Trauma, Nervous System

STUDY DESIGN:
Intervention Model Description: From the patients who came for consultation between 2015 and 2020, subjects have been recruited by mail for the Coronaltitude study from the 1st of March (2021) on. Subjects have been asked if they have suffered COVID19 in the 12 months before inclusion, during whichever wave, attested by a positive PCR, positive serology test or positive chest CT scan. Both patients answering positively and those answering negatively on the latter question have been included in the study. All included subjects, divided into those having suffered COVID19 (COVID+ group) and those having stayed free of COVID19 (control group), will retake an altitude mountain consultation.
Masking Description: All subjects, whether partaking in the COVID+ group or control group, got the same intervention. As such, the 'intervention' rather is the having undergone COVID19 or not. Involving sanitary reasons surrounding the COVID pandemic, a lack of communication concerning the COVID diagnosis between and to any party would have led to unnecessary health endangerment of concerned parties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID+ group (Experimental): As the performance of the Richalet test is done by both arms, the intervention rather is the having undergone COVID19.
  Interventions: Biological: COVID19
- Control group / COVID- group (No Intervention): Performance of the Richalet test is done by both arms, the control in this study here is the having stayed clear of COVID19.

INTERVENTIONS:
Biological: COVID19 — Intervention in experimental group (COVID+ group) is the disease itself, compared to the control group (COVID- group). At inclusion, subjects have been asked if they have suffered COVID19 in the 12 months before inclusion, during whichever wave, attested by a positive PCR, positive serology test or positive chest CT scan.
  Moreover, the Richalet test is a cardiorespiratory exercise test on an ergocycle (an electrically braked cycloergometer), whilst continuous measurement by a 12-lead ECG, a blood pressure cuff, a metabograph and an ear pulse oximeter. This, to assess cardiac response, ventilatory response and relevant metabolic parameters (CF, RR, SpO2, volume, BP). Subjects breathes through a mask connected to a gas mixer, which provides a gas mixture with 11,5% oxygen (corresponding to ambient air at an altitude of 4800m) in the hypoxia phases.
  Other Names: SARS-CoV-2; Covid; severe acute respiratory syndrome coronavirus 2
  Arms: COVID+ group

SUMMARY:
In this study, the investigators will examine the extent to which having suffered coronavirus disease 2019 (COVID19) impacts one's sensibility to hypoxia by means of the 'Richalet test'. The aim of the study is to formulate recommendations for advice in altitude mountain medicine for patients having suffered COVID19. To determine any eventual changes in response to hypoxia, performances by participants having suffered COVID-19 and participants having stayed free of COVID-19 will be both compared intra-individually with previous performances (pre-COVID-19 pandemic) and between both groups of subjects. The investigators hypothesize that patients having suffered COVID19 might perform differently on the cardiopulmonary exercise test compared to before the illness. Based on recent research on COVID19 pathophysiology and -patient follow-up, it might be expected that COVID19 alters the response to hypoxia, thus influencing one's acclimatization capabilities at high altitude, albeit reversibly and/or temporarily.

Different alterations of response to hypoxia could be observed. The virus causing COVID19, the "severe acute respiratory syndrome coronavirus 2" (SARS-CoV-2), has the potential to significantly damage the nervous system and to affect cardiorespiratory functions. If SARS-CoV-2 does, similarly to MERS and SARS, induce cardiorespiratory and neurological dysfunction, then COVID19 patients may have impaired hypoxia response after infection and perform worse on the 'Richalet test' in comparison to before the illness.

Conversely, reports of high prevalence of dyspnea in patients up to 3 months after SARS-CoV-2 infection, might indicate infection-induced degenerative changes in the carotid bodies, which might lead to sensibilization of the peripheral chemoreceptors to impaired oxygenation. Possibly similar to the impact of aging and smoking on the cardiorespiratory response to hypoxia, this phenomenon of sensibilization could entail an increased hypoxic response in patients having suffered COVID-19. Accordingly, patients might perform better on the 'Richalet test' post-COVID-19 than they did before.

DETAILED DESCRIPTION:
In this study, the focus will be on the portion of COVID-19 survivors which contemplates to travel to and (temporarily) reside in high altitude regions (>2500m). It is well known that as altitude increases, the barometric pressure falls, proportionally paralleled by a decreasing partial pressure of oxygen. At high altitude, this leads to a condition which is referred to as a hypobaric hypoxic environment. The dramatic drop in partial pressure of inspired oxygen and subsequent reduction in arterial partial pressure of oxygen implicates significant adjustments for the human body to survive at high altitude. In order to study the possible long-term effects of COVID-19 on oxygen transport physiology in these patients, the investigators will focus on the eventual cardiorespiratory and neurological consequences of SARS-CoV-2 infection and relate them to the physiological demands placed on the body by hypoxia at high altitude. This case-control study will be conducted by means of the 'Richalet Test', a hypoxia cardiorespiratory exercise test which has been validated for mountain medicine consultations to detect patients at risk of developing an inadequate response to hypoxia at high altitude. From the patients who came for consultation between 2015 and 2020, participants have been recruited by mail for the Coronaltitude study. All included participants, divided into those having suffered COVID-19 (COVID+ group) and those having stayed free of COVID-19 (control group), will retake an altitude mountain consultation. Results will be compared in between and within both groups with previous performances to determine if the response to hypoxia has changed in people having undergone COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Subject having suffered COVID19 in the 12 months before inclusion, attested by a positive PCR, positive serology test or positive chest CT scan. (COVID+ group).
* Subject having stayed clear of COVID19 (COVID-/control group).
* Subject having been well informed and having provided written informed consent before participation.
* Subject covered by social security of some sort.
* Subject with an oxygen saturation of SpO2 > 95% in ambient air on day of Richalet test performance.
* Subject presenting with no symptoms of COVID19 (anymore) on the day of the experiment.
* Subject having already performed the Richalet hypoxia exercise test as part of the altitude mountain consultation in the years 2015 to 2019 in any of the 13 hospital centers participating at the study.

Exclusion Criteria:

* Subject with a history of respiratory, cardiovascular, neuromuscular, metabolic or renal pathologies.
* Subject with a history of psychiatric or behavioral disorder.
* Subject covered by L1121-5 to L1121-8 sections of the Public Health regulations (Code de la Santé Publique).
* Subject under guardian- or curatorship.
* Subject without social insurance.
* Subjet under the age of 18.
* Subject refusing to participate in the study.
* Subject diagnosed with an infection by a pathogen other than SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
desaturation induced by hypoxia at exercise (∆SaO2) | Continuous measuring during the entirety of the hypoxia exercise test over a period of time of around 30 min with cornerstone measurements every 4 min.
  ∆SaO2, HCRe and HVRe are considered to be indirect measurements of the chemosensitivity and response to hypoxia. HCRe and HVRe are calculated from the ratio of respective increased parameters (CF and RR) over the decrease in arterial oxygen saturation measured in 5 consecutive phases of the hypoxic exercise test.
hypoxic cardiac response at exercise (HCRe) | Continuous measuring during the entirety of the hypoxia exercise test over a period of time of around 30 min with cornerstone measurements every 4 min.
  See description outcome 1
hypoxic ventilatory response at exercise (HVRe) | Continuous measuring during the entirety of the hypoxia exercise test over a period of time of around 30 min with cornerstone measurements every 4 min.
  see description outcome 1

SECONDARY OUTCOMES:
SHAI prediction score | Assessment over a period of time of a common mountain consultation - around half a day.
  Calculated by means of obtained results of the Richalet test combined with normalized answers to the altitude mountain consultation questionnaires. In turn, normalized SHAI scores are also compared within and in between both groups in order to evaluate the eventual impact of having suffered COVID19 one one's susceptibility to develop SHAI symptoms. Assessment after each subject has performed the Richalet test - using the by the multiSHAI study validated computation of the SHAI score to define the individual susceptibility to Severe High Altitude Illness (SHAI).

CONTACTS AND LOCATIONS:
Overall Officials: François Lecoq-Jammes, Dr., Principal Investigator — study coordinator
Locations (1):
- Institut de Formation et de Recherche en Médecine de Montagne (IFREMMONT), Chamonix, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Richalet JP, Pillard F, LE Moal D, Riviere D, Oriol P, Poussel M, Chenuel B, Doutreleau S, Verges S, Demanez S, Vergnion M, Boulet JM, Douard H, Dupre M, Mesland O, Remetter R, Lonsdorfer-Wolf E, Frey A, Vilcoq L, Nedelec Jaffuel A, Debeaumont D, Duperrex G, Lecoq F, Hedon C, Hayot M, Giardini G, Lhuissier FJ. Validation of a Score for the Detection of Subjects with High Risk for Severe High-Altitude Illness. Med Sci Sports Exerc. 2021 Jun 1;53(6):1294-1302. doi: 10.1249/MSS.0000000000002586. PMID 33433150
- [Background] Richalet JP, Canoui-Poitrine F. Pro: hypoxic cardiopulmonary exercise testing identifies subjects at risk for severe high altitude illnesses. High Alt Med Biol. 2014 Sep;15(3):315-7. doi: 10.1089/ham.2014.1032. No abstract available. PMID 25251925
- [Background] Cao Y, Liu X, Xiong L, Cai K. Imaging and clinical features of patients with 2019 novel coronavirus SARS-CoV-2: A systematic review and meta-analysis. J Med Virol. 2020 Sep;92(9):1449-1459. doi: 10.1002/jmv.25822. Epub 2020 Apr 10. PMID 32242947
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Higgins V, Sohaei D, Diamandis EP, Prassas I. COVID-19: from an acute to chronic disease? Potential long-term health consequences. Crit Rev Clin Lab Sci. 2021 Aug;58(5):297-310. doi: 10.1080/10408363.2020.1860895. Epub 2020 Dec 21. PMID 33347790
- [Background] Luks AM, Grissom CK. Return to High Altitude After Recovery from Coronavirus Disease 2019. High Alt Med Biol. 2021 Jun;22(2):119-127. doi: 10.1089/ham.2021.0049. Epub 2021 May 11. PMID 33978479
- [Background] Canoui-Poitrine F, Veerabudun K, Larmignat P, Letournel M, Bastuji-Garin S, Richalet JP. Risk prediction score for severe high altitude illness: a cohort study. PLoS One. 2014 Jul 28;9(7):e100642. doi: 10.1371/journal.pone.0100642. eCollection 2014. PMID 25068815
- [Background] Coustet B, Lhuissier FJ, Vincent R, Richalet JP. Electrocardiographic changes during exercise in acute hypoxia and susceptibility to severe high-altitude illnesses. Circulation. 2015 Mar 3;131(9):786-94. doi: 10.1161/CIRCULATIONAHA.114.013144. Epub 2015 Jan 5. PMID 25561515
- [Background] Richalet JP, Larmignat P, Poitrine E, Letournel M, Canoui-Poitrine F. Physiological risk factors for severe high-altitude illness: a prospective cohort study. Am J Respir Crit Care Med. 2012 Jan 15;185(2):192-8. doi: 10.1164/rccm.201108-1396OC. Epub 2011 Oct 27. PMID 22071330
- [Background] Algahtani H, Subahi A, Shirah B. Neurological Complications of Middle East Respiratory Syndrome Coronavirus: A Report of Two Cases and Review of the Literature. Case Rep Neurol Med. 2016;2016:3502683. doi: 10.1155/2016/3502683. Epub 2016 Apr 28. PMID 27239356
- [Background] Desforges M, Le Coupanec A, Dubeau P, Bourgouin A, Lajoie L, Dube M, Talbot PJ. Human Coronaviruses and Other Respiratory Viruses: Underestimated Opportunistic Pathogens of the Central Nervous System? Viruses. 2019 Dec 20;12(1):14. doi: 10.3390/v12010014. PMID 31861926
- [Background] Li YC, Bai WZ, Hashikawa T. The neuroinvasive potential of SARS-CoV2 may play a role in the respiratory failure of COVID-19 patients. J Med Virol. 2020 Jun;92(6):552-555. doi: 10.1002/jmv.25728. Epub 2020 Mar 11. PMID 32104915
- [Background] Montalvan V, Lee J, Bueso T, De Toledo J, Rivas K. Neurological manifestations of COVID-19 and other coronavirus infections: A systematic review. Clin Neurol Neurosurg. 2020 Jul;194:105921. doi: 10.1016/j.clineuro.2020.105921. Epub 2020 May 15. PMID 32422545
- [Background] Ellul MA, Benjamin L, Singh B, Lant S, Michael BD, Easton A, Kneen R, Defres S, Sejvar J, Solomon T. Neurological associations of COVID-19. Lancet Neurol. 2020 Sep;19(9):767-783. doi: 10.1016/S1474-4422(20)30221-0. Epub 2020 Jul 2. PMID 32622375
- [Background] Salehi S, Reddy S, Gholamrezanezhad A. Long-term Pulmonary Consequences of Coronavirus Disease 2019 (COVID-19): What We Know and What to Expect. J Thorac Imaging. 2020 Jul;35(4):W87-W89. doi: 10.1097/RTI.0000000000000534. No abstract available. PMID 32404798
- [Background] Huang Y, Tan C, Wu J, Chen M, Wang Z, Luo L, Zhou X, Liu X, Huang X, Yuan S, Chen C, Gao F, Huang J, Shan H, Liu J. Impact of coronavirus disease 2019 on pulmonary function in early convalescence phase. Respir Res. 2020 Jun 29;21(1):163. doi: 10.1186/s12931-020-01429-6. PMID 32600344
- [Background] Zhao YM, Shang YM, Song WB, Li QQ, Xie H, Xu QF, Jia JL, Li LM, Mao HL, Zhou XM, Luo H, Gao YF, Xu AG. Follow-up study of the pulmonary function and related physiological characteristics of COVID-19 survivors three months after recovery. EClinicalMedicine. 2020 Aug;25:100463. doi: 10.1016/j.eclinm.2020.100463. Epub 2020 Jul 15. PMID 32838236
- [Background] Zubieta-Calleja G, Zubieta-DeUrioste N. Pneumolysis and "Silent Hypoxemia" in COVID-19. Indian J Clin Biochem. 2021 Jan;36(1):112-116. doi: 10.1007/s12291-020-00935-0. Epub 2020 Nov 9. PMID 33191989
- [Background] Zubieta-Calleja G, Zubieta-DeUrioste N, Venkatesh T, Das KK, Soliz J. COVID-19 and Pneumolysis Simulating Extreme High-altitude Exposure with Altered Oxygen Transport Physiology; Multiple Diseases, and Scarce Need of Ventilators: Andean Condor's-eye-view. Rev Recent Clin Trials. 2020;15(4):347-359. doi: 10.2174/1574887115666200925141108. PMID 32981508
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Nouri-Vaskeh M, Sharifi A, Khalili N, Zand R, Sharifi A. Dyspneic and non-dyspneic (silent) hypoxemia in COVID-19: Possible neurological mechanism. Clin Neurol Neurosurg. 2020 Nov;198:106217. doi: 10.1016/j.clineuro.2020.106217. Epub 2020 Sep 9. PMID 32947193
- [Background] Couzin-Frankel J. The mystery of the pandemic's 'happy hypoxia'. Science. 2020 May 1;368(6490):455-456. doi: 10.1126/science.368.6490.455. No abstract available. PMID 32355007
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Goertz YMJ, Van Herck M, Delbressine JM, Vaes AW, Meys R, Machado FVC, Houben-Wilke S, Burtin C, Posthuma R, Franssen FME, van Loon N, Hajian B, Spies Y, Vijlbrief H, van 't Hul AJ, Janssen DJA, Spruit MA. Persistent symptoms 3 months after a SARS-CoV-2 infection: the post-COVID-19 syndrome? ERJ Open Res. 2020 Oct 26;6(4):00542-2020. doi: 10.1183/23120541.00542-2020. eCollection 2020 Oct. PMID 33257910
- [Background] Richalet JP, Lhuissier FJ. Aging, Tolerance to High Altitude, and Cardiorespiratory Response to Hypoxia. High Alt Med Biol. 2015 Jun;16(2):117-24. doi: 10.1089/ham.2015.0030. Epub 2015 May 6. PMID 25946570
- [Background] Hackett PH, Roach RC. High-altitude illness. N Engl J Med. 2001 Jul 12;345(2):107-14. doi: 10.1056/NEJM200107123450206. No abstract available. PMID 11450659
- [Background] Neubauer JA, Melton JE, Edelman NH. Modulation of respiration during brain hypoxia. J Appl Physiol (1985). 1990 Feb;68(2):441-51. doi: 10.1152/jappl.1990.68.2.441. PMID 2180894
- [Background] Bartsch P, Swenson ER. Clinical practice: Acute high-altitude illnesses. N Engl J Med. 2013 Jun 13;368(24):2294-302. doi: 10.1056/NEJMcp1214870. PMID 23758234
- [Background] Lovis A, Gabus V, Daucourt C, De Riedmatten M, Sartori C. [Hypoxic tests and prediction of high altitude illnesses]. Rev Med Suisse. 2019 May 1;15(649):917-922. French. PMID 31050239
- [Background] Hohenhaus E, Paul A, McCullough RE, Kucherer H, Bartsch P. Ventilatory and pulmonary vascular response to hypoxia and susceptibility to high altitude pulmonary oedema. Eur Respir J. 1995 Nov;8(11):1825-33. doi: 10.1183/09031936.95.08111825. PMID 8620946
- [Background] Schoene RB, Roach RC, Hackett PH, Sutton JR, Cymerman A, Houston CS. Operation Everest II: ventilatory adaptation during gradual decompression to extreme altitude. Med Sci Sports Exerc. 1990 Dec;22(6):804-10. PMID 2287258
- [Background] Hackett PH. The cerebral etiology of high-altitude cerebral edema and acute mountain sickness. Wilderness Environ Med. 1999 Summer;10(2):97-109. doi: 10.1580/1080-6032(1999)010[0097:tceoha]2.3.co;2. PMID 10442158
- [Background] Basnyat B, Cumbo TA, Edelman R. Infections at high altitude. Clin Infect Dis. 2001 Dec 1;33(11):1887-91. doi: 10.1086/324163. Epub 2001 Oct 19. PMID 11668431
- [Background] Song TT, Bi YH, Gao YQ, Huang R, Hao K, Xu G, Tang JW, Ma ZQ, Kong FP, Coote JH, Chen XQ, Du JZ. Systemic pro-inflammatory response facilitates the development of cerebral edema during short hypoxia. J Neuroinflammation. 2016 Mar 11;13(1):63. doi: 10.1186/s12974-016-0528-4. PMID 26968975
- [Derived] Louis A, Propper C, Savina Y, Tanne C, Duperrex G, Robach P, Zellner P, Doutreleau S, Boulet JM, Frey A, Pillard F, Pistea C, Poussel M, Thuet T, Richalet JP, Lecoq-Jammes F. The Impact of COVID-19 on the Response to Hypoxia. High Alt Med Biol. 2023 Dec;24(4):321-328. doi: 10.1089/ham.2022.0156. Epub 2023 Oct 16. PMID 37843910